CLINICAL TRIAL: NCT03864237
Title: Correcting Exaggerated Drinking Norms With a Mobile Message Delivery System
Brief Title: Text-based Alcohol Prevention for First Year College Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Responsible Party: Principal Investigator, Kate Carey, Professor, Brown University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R21AA024771 (NIH)
Record Dates: First submitted 2018-09-11; First posted 2019-03-06 (Actual); Results first posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: College Drinking
Keywords: alcohol abuse; college students; preventive programs; text messages
MeSH Terms: conditions — Alcohol Drinking in College; Alcoholism | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alcohol texts (Experimental): Participants assigned to this arm will receive a text message each day for 10 weeks, containing factual information about campus drinking norms.
  Interventions: Behavioral: Alcohol texts
- Attention control (Placebo Comparator): Participants assigned to this arm will receive a text message each day for 10 weeks, containing "this day in history" facts.
  Interventions: Behavioral: Attention control

INTERVENTIONS:
Behavioral: Alcohol texts — A text message each day for 10 weeks, containing factual information about campus drinking norms.
  Arms: Alcohol texts
Behavioral: Attention control — A text message each day for 10 weeks, containing "this day in history" facts.
  Arms: Attention control

SUMMARY:
This project aims to combat excessive perceived norms that contribute to high volume drinking by young adults, which adversely affects health and academic achievement. Campus-specific survey data will be used to craft accurate, pro-moderation campus norms, and deliver them to first-year students via daily text messages during the first semester of college. It is predicted that those receiving regular exposure to pro-moderation drinking norms will reduce their alcohol consumption and consequences, relative to students who receive non-alcohol-related control texts. This preliminary evaluation uses a novel method of delivering drinking norms and will lay the groundwork for future efforts to scale up this novel alcohol misuse prevention approach.

DETAILED DESCRIPTION:
Using mobile technology that most students already have in their pockets, this study evaluates a novel use of text messages to change campus drinking norms. The aim is to correct exaggerated perceptions of drinking norms, and thereby reduce excessive drinking, by delivering daily text messages representing accurate, campus-specific, pro-moderation descriptive norms (what others do) and injunctive norms (what others approve of). It is predicted that with repeated exposure over time, this information will compete with other sources of normative information to which students are exposed during their first year of college. This exploratory study is designed to develop and refine message content and to pilot test the delivery methods.

First year students (N=120) who are underage but report risky drinking (>4/day or >14/week for men; >3/day or >7/week for women) will be randomly assigned to two conditions differing by text content: alcohol norms or attention control. All will receive daily text messages throughout 10 weeks in the first semester of college. Process measures, 3-month post-test, and 3-month follow-up assessments will yield feasibility, acceptability, and preliminary outcome data to inform future larger scale randomized trials. Specifically, baseline, post-test, and 3-month follow-up assessments will allow us to test the hypotheses that the corrective norms intervention will reduce (a) perceived descriptive and injunctive norms, (b) drinking behavior (including high-volume drinking and risky consumption practices), and (c) alcohol-related consequences, and increase (d) protective behavioral strategies, relative to the control condition.

At the end of this project the investigative team will have gathered data on both descriptive and injunctive norms on a range of drinking behaviors to identify topics in need of corrective normative feedback, refined the structure and content of the text messages, and pilot tested the text-delivered intervention in a small scale randomized controlled trial (RCT). The proposed research will provide evidence of feasibility and efficacy of a text-based alcohol norms intervention for reducing excessive drinking among first-year students.

ELIGIBILITY:
Inclusion Criteria:

* 18-20 years of age
* enrolled as a first-year undergraduate student
* past month risky drinking
* possession of a mobile phone with text message capacity
* use text messaging at least weekly

Exclusion Criteria:

* currently engaged in alcohol treatment or in need of treatment (AUDIT score 20 or higher)

Ages: 18 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 121 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Brown University, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
After all data have been collected and results of the study have been published, de-identified data will be made available to other qualified investigators upon request. The request will be evaluated by the investigators to ensure that it meets reasonable expectations of scientific integrity.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: within one year of study completion, for up to 3 years
Access Criteria: to be determined

REFERENCES:
- [Derived] Carey KB, Merrill JE, Boyle HK, Barnett NP. Correcting exaggerated drinking norms with a mobile message delivery system: Selective prevention with heavy-drinking first-year college students. Psychol Addict Behav. 2020 May;34(3):454-464. doi: 10.1037/adb0000566. Epub 2020 Mar 2. PMID 32118463

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligibility was determined via an online screening survey distributed by email during the first few weeks of the fall 2018 semester to all first-year students enrolled at the university. Eligible participants were directed to an online consent form and then emailed a link to an online baseline survey.
Period: Overall Study
Arm/Group | Alcohol Texts | Attention Control
Started | 61 | 60
Completed | 61 | 60
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alcohol Texts | Attention Control | Total
Number analyzed (Participants) | 61 | 60 | 121
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 61 | 60 | 121
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.5 (0.36) | 18.1 (0.30) | 18.12 (0.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 30 | 61
  Male | 30 | 30 | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 9 | 19
  Not Hispanic or Latino | 51 | 51 | 102
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 13 | 9 | 22
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 5 | 10
  White | 32 | 38 | 70
  More than one race | 3 | 4 | 7
  Unknown or Not Reported | 8 | 4 | 12
Region of Enrollment [Number; unit: participants]
  United States | 61 | 60 | 121
Drinks per week [Mean (Standard Deviation); unit: drinks per week] — Drinks per week as measured by the Daily Drinking Questionnaire. Drinks per week is determined by counting up the typical number of drinks entered on each of the 7 days of the week, to get a sum.
  drinks per week | 11.42 (6.15) | 12.79 (7.13) | 12.10 (6.66)
Alcohol-related consequences [Mean (Standard Deviation); unit: consequences] — Alcohol-related consequences are a count of the number of items endorsed on the 24-item Brief Young Adult Alcohol Consequences Questionnaire. The range is 0-24, and represents the number of consequences experienced over the last month.
  consequences | 4.95 (2.87) | 4.35 (2.67) | 4.65 (2.78)

OUTCOME MEASURES:

1. Primary Outcome: Drinks Per Week as Assessed by the Daily Drinking Questionnaire
Description: Sum of standard drinks consumed on each day in a typical week over the past 30 days; scores can be as low as zero but there is no upper limit as they are counts of drinks
Time Frame: Assessed over prior 30 days at 3 month follow-up
Measure: Mean (Standard Deviation); unit: drinks per week
Arm/Group | Alcohol Texts | Attention Control
Number analyzed (Participants) | 56 | 58
drinks per week | 9.55 (6.02) | 10.87 (6.24)
Statistical Analysis 1: Comparison: Alcohol Texts vs Attention Control; Test type: Superiority; p = 0.568, Regression, Linear; Regression controls for baseline value of outcome and sex to determine pre-post change in the outcome as a function of condition; beta coefficient for condition = 0.53, 95% CI 2-sided [-1.31 to 2.37], Standard Error of Mean 0.93

2. Primary Outcome: Alcohol-related Consequences as Assessed by the Brief Young Adult Alcohol Consequences Questionnaire
Description: The total number of alcohol-related consequences experienced over the past 30 days is measured by the Brief Young Adult Alcohol Consequences Questionnaire (BYAACQ), which is a checklist of 24 items; scores range from 0-24; higher numbers of items endorsed indicate more problems experienced in the past 30 days
Time Frame: Assessed over prior 30 days at 3 month follow-up
Measure: Mean (Standard Deviation); unit: consequences
Arm/Group | Alcohol Texts | Attention Control
Number analyzed (Participants) | 57 | 57
consequences | 4.44 (3.52) | 5.32 (4.08)
Statistical Analysis 1: Comparison: Alcohol Texts vs Attention Control; Test type: Superiority; p = 0.077, Regression, Linear; beta coefficient for condition = 1.22, 95% CI 2-sided [-0.13 to 2.59], Standard Error of Mean 0.69

3. Secondary Outcome: Protective Behavioral Strategies as Assessed by the Strategies Questionnaire - Alternative Sub Scale
Description: self-reported frequency of using strategies to moderate drinking as reported on the Strategy Questionnaire; the Strategy Questionnaire has 3 sub scales including Selective Avoidance (0-70), Strategies While Drinking (0-100), and Alternatives to Drinking (0-40) and higher sub scale scores indicate more frequent use of those strategies
Time Frame: Assessed over prior 30 days at 3 month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Alcohol Texts | Attention Control
Number analyzed (Participants) | 57 | 57
score on a scale | 14.54 (5.75) | 13.53 (8.15)
Statistical Analysis 1: Comparison: Alcohol Texts vs Attention Control; Test type: Superiority; p = 0.30, Regression, Linear; beta coefficient for condition = -1.21, 95% CI 2-sided [-3.52 to 1.11], Standard Error of Mean 1.17

4. Secondary Outcome: Perceived Descriptive Drinking Norms as Assessed by the Drinking Norms Rating Form
Description: perceived descriptive norms are assessed using a variation on the Drinking Norms Rating Form, which asks respondents to estimate the number of standard drinks consumed by other students on campus for each day in a typical week in the past 30 days; daily estimates are summed to yield perceived number of drinks per week for student peers; range of scores can go from zero to no upper limit
Time Frame: Assessed over prior 30 days at 3 month follow-up
Measure: Mean (Standard Deviation); unit: drinks per week
Arm/Group | Alcohol Texts | Attention Control
Number analyzed (Participants) | 57 | 57
drinks per week | 11.46 (6.43) | 12.74 (6.87)
Statistical Analysis 1: Comparison: Alcohol Texts vs Attention Control; Test type: Superiority; p = 0.44, Regression, Linear; beta coefficient for condition = 0.84, 95% CI 2-sided [-1.31 to 3.0], Standard Error of Mean 1.09

5. Secondary Outcome: Perceived Injunctive Drinking Norms as Assessed by an Adaptation of the Drinking Norms Rating Form
Description: perceived injunctive norms are assessed using the Krieger et al. (2016) adaptation of the Drinking Norms Rating Form, which asks respondents to estimate the how many standard drinks is deemed acceptable by other students on campus to drink on each day in a typical week in the past 30 days; estimates are summed to yield number of drinks per week approved of by student peers; the scores can range from zero to no upper limit
Time Frame: Assessed over prior 30 days at 3 month follow-up
Measure: Mean (Standard Deviation); unit: drinks per week
Arm/Group | Alcohol Texts | Attention Control
Number analyzed (Participants) | 57 | 57
drinks per week | 15.72 (8.79) | 16 (8.70)
Statistical Analysis 1: Comparison: Alcohol Texts vs Attention Control; Test type: Superiority; p = 0.845, Regression, Linear; Beta coefficient for condition = -0.25, 95% CI 2-sided [-2.81 to 2.30], Standard Error of Mean 1.29

6. Secondary Outcome: Protective Behavioral Strategies as Assessed by the Strategies Questionnaire - Selective Avoidance Sub Scale
Description: as for outcome 3
Time Frame: Assessed over prior 30 days at 3 month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Alcohol Texts | Attention Control
Number analyzed (Participants) | 53 | 54
score on a scale | 5.9 (6.66) | 5.67 (5.64)
Statistical Analysis 1: Comparison: Alcohol Texts vs Attention Control; Test type: Superiority; p = 0.77, Regression, Linear; Beta coefficient for condition = 0.30, 95% CI 2-sided [-1.72 to 2.31], Standard Error of Mean 1.01

7. Secondary Outcome: Protective Behavioral Strategies as Assessed by the Strategies Questionnaire - Strategies Sub Scale
Description: as for outcome 3
Time Frame: Assessed over prior 30 days at 3 month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Alcohol Texts | Attention Control
Number analyzed (Participants) | 53 | 54
score on a scale | 12.90 (7.75) | 13.51 (8.16)
Statistical Analysis 1: Comparison: Alcohol Texts vs Attention Control; Test type: Superiority; p = 0.21, Regression, Linear; Beta coefficient for condition = 1.77, 95% CI 2-sided [-1.0 to 4.54], Standard Error of Mean 1.40

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Alcohol Texts | Attention Control
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/60
Other Adverse Events (participants affected / at risk) | 0/61 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-09-21): https://cdn.clinicaltrials.gov/large-docs/37/NCT03864237/Prot_SAP_000.pdf
  • Informed Consent Form (2018-08-06): https://cdn.clinicaltrials.gov/large-docs/37/NCT03864237/ICF_001.pdf